CLINICAL TRIAL: NCT02467491
Title: A New Adaptive Physical Activity Technology in Older Adults (Jintronix)
Brief Title: A New Adaptive Physical Activity Technology in Older Adults
Acronym: Jintronix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IRB201500368
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Aging
Keywords: Exercise; Technology; Aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Activity group (Other): All the participants enrolled in the study will be part of the physical activity group in which they will perform a scheduled exercise program for 4 weeks using a new physical activity technology called Jintronix.
  Interventions: Device: Jintronix

INTERVENTIONS:
Device: Jintronix — The participants will perform light exercises using the Jintronix software. Jintronix is an easy-to-use virtual physical activity platform designed for physical and occupational therapy. It combines common exercise movements, virtual games and motion sensing cameras to offer a fun and effective tool for physical activity.

SUMMARY:
The purpose of this study is to explore the feasibility and acceptability of a new physical activity technology (Jintronix) based on TV screen, virtual games and motion sensing cameras among pre-disabled older adults.

DETAILED DESCRIPTION:
A total of 12 older adults will be recruited in the Oak Hammock residential community to participate in a physical activity program using a new technology called Jintronix. Jintronix is an easy-to-use virtual physical activity platform designed for physical and occupational therapy. It combines common exercise movements, virtual games and motion sensing cameras to offer a fun and effective tool for physical activity. The exercises will be performed by each participant autonomously in the living room of the residential community following a specific schedule. The duration of the exercise program will be of 30 minutes for two days a week for a total of four weeks. The participants will be trained prior the beginning of the program in order to enter autonomously in the Jintronix platform and perform the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and older
* Pre-disabled status evidenced by: 6 ≤ score ≤ 9 on the Short Physical Performance Battery test.
* Willingness to participate in all study procedures.

Exclusion Criteria:

* Failure to provide informed consent
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Significant cognitive impairment, defined as a known diagnosis of dementia or a short portable mental status questionnaire score > 2 errors
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment, which would preclude completion of the assessments and/or exercise program
* Other significant co-morbid diseases that would prevent participation in exercise
* Planning to move out of the area during the study timeframe

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Valiani, MD, Principal Investigator — University of Florida
Locations (1):
- Oak Hammock at University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants signed the informed consent, but only 12 participants started and completed the exercise intervention
Period: Overall Study
Arm/Group | Physical Activity Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Older adults living in the residential community Oak Hammock at University of Florida
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.5 (2.9)
Short Physical Performance Battery score (SPPB) [Mean (Standard Deviation); unit: units on a scale] — The SPPB is a common measure of physical performance in older adults. The test is comprised of timed measures of standing balance in three positions (side by side position, semi tandem position, tandem position), walking speed over 4 meters, and time to stand up and sit down 5 times in a chair, as quickly as possible. Each of the 3 performance measures are assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the test. A summary score was created by adding each performance score and ranges from 0-12.
  units on a scale | 8.2 (1.2)
Rapid Assessment of Physical Activity (RAPA) score [Mean (Standard Deviation); unit: units on a scale] — The Rapid Assessment of Physical Activity (RAPA) questionnaire is a questionnaire made of 7 questions that ask about the amount and intensity of physical activity during the week. Minimum score is 0 and maximum score is 7 as described below:
  Sedentary: score 1 Under-active: score 2 Under-active regular-light activities: score 3 Under-active regular: score 4 or 5 Active: score 6 or 7
  units on a scale | 4.08 (1.44)
Short Portable Mental Status Questionnaire score [Mean (Standard Deviation); unit: units on a scale] — The Short Portable Mental Status Questionnaire is made of 8 questions which explore the cognitive function of the subject. Possible scores range from 0 to 8 with lower scores indicating better cognitive function.
  units on a scale | 0.08 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Movements' Total Average Score
Description: The quality of movements' score is a measure of feasibility. The quality of movement's score is automatically calculated by Jintronix for each participant at the end of the intervention program with Jintronix.
  A quality of movement's score of 100% means that the participant performed the exercise perfectly.
  To calculate the quality of movements' total average score for the Group (made of 12 participants), we summed the quality of movements' score for each participants and divided it for 12. We expected to find a total average quality movements' score>80% in order to say that Jintronix was feasible.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of quality of movements
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
percentage of quality of movements | 87 (10)

2. Primary Outcome: Total Average Time in Performing Exercises With Jintronix.
Description: Each participant has to perform the exercise program with Jintronix for 30 minutes per session, for 2 times/week for a total of 4 weeks.
  This means that each participant has to be able to perform a maximum of 240 minutes of exercises for 4 weeks.
  Jintronix calculated automatically the time (minutes) in performing the exercises for each participant at the end of the 4 weeks of intervention.
  As a measure of acceptability we calculated the total average time in performing the exercises for the 12 participants for 4 weeks by summing the minutes in performing the exercises for each participants for 4 week and dividing it for 12.
  We expected to find an average total time in performing the exercises for 12 participants > 192 minutes (3.2 hours) out of a total of 240 minutes (4 hours) in order to say that Jintronix was acceptable.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
minutes | 207.5 (32.51)

3. Primary Outcome: Global Difficulty Score
Description: The global difficulty score was another measure of acceptability.
  The global difficulty score will be derived from each participant's answer to the second question of a 9-item feasibility questionnaire. The second question of the questionnaire is :"How difficult did you find the Jintronix?", participants' answer may be:
  * Very difficult (3 point)
  * Quite difficult (2 points)
  * Not at all (1 points)
  * No difficulty (0 points). This means that the global difficulty score for 12 participants may range from 0 (no difficult) to 36 (very difficult).
  We expected to find a global difficulty score < to 15 in order to say that Jintronix was acceptable.
Time Frame: 4 weeks
Measure: Number; unit: units on a scale
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
units on a scale | 13

4. Primary Outcome: Global Appreciation Score
Description: The global appreciation score is a measure of feasibility.
  This score will be derived from each participant's answer to the first question of a 9-item acceptability questionnaire. The second question of the questionnaire is :"How much did you like Jintronix?", participants' answer may be:
  * I didn't like it (0 point)
  * A little (1 points)
  * Moderate (2 points)
  * A lot (3 points). The global appreciation score is the sum of the points obtained by each participants.
  The global appreciation score for 12 participants may range from 0 (no appreciation) to 36 (a lot of appreciation).
  In order to say that Jintronix is feasible we expected a global appreciation score for 12 participant after 4 weeks of intervention to be > 24.
Time Frame: 4 weeks
Measure: Number; unit: units on a scale
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
units on a scale | 33

5. Secondary Outcome: Change From Baseline to 4 Weeks in the Short Physical Performance Battery Test
Description: Physical performance will be assessed using the Short Physical Performance Battery test (SPPB). The score for this test is 0 meaning the worst performance to 12 meaning the best performance.
Time Frame: Change in baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
units on a scale | 0.67 (0.98)
Statistical Analysis 1: Comparison: Physical Activity Group; The Short Physical Performance Battery (SPPB) score at baseline was compared with the SPPB scored after 4 weeks of physical activity intervention with a paired t-test; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

6. Secondary Outcome: Change From 4 Weeks (End of Intervention) to 3 Months After the End of the Intervention in the Short Physical Performance Battery Test
Description: as for outcome 5
Time Frame: Change in 4 weeks to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Group
Number analyzed (Participants) | 12
units on a scale | 0.42 (0.51)
Statistical Analysis 1: Comparison: Physical Activity Group; The Short Physical Performance Battery (SPPB) score after 4 weeks of physical activity intervention was compared with the SPPB score after 2 to 3 months from the completion of the physical activity intervention with a paired t-test; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Physical Activity Group
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No